CLINICAL TRIAL: NCT02568254
Title: Evaluation of Three Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CR-5735
Record Dates: First submitted 2015-09-22; First posted 2015-10-05 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Lens 1/ Lens 2/ Lens 3 (Active Comparator): Each subject will be randomly assigned to one of six unique sequences. Subjects randomized to this sequence will first wear Lens 1 (etafilcon A), then wear Lens 2 (nelfilcon A) second and then wear Lens 3 (nesofilcon A) third.
  Interventions: Device: Lens 1 (etafilcon A); Device: Lens 2 (nelfilcon A); Device: Lens 3 (nesofilcon A)
- Lens 1 / Lens 3 / Lens 2 (Active Comparator): Each subject will be randomly assigned to one of six unique sequences. Subjects randomized to this sequence will first wear Lens 1 (etafilcon A), then wear Lens 3 (nesofilcon A) second and then wear Lens 2 (nelfilcon A) third.
  Interventions: Device: Lens 1 (etafilcon A); Device: Lens 2 (nelfilcon A); Device: Lens 3 (nesofilcon A)
- Lens 2/ Lens 3/ Lens 1 (Active Comparator): Each subject will be randomly assigned to one of six unique sequences. Subjects randomized to this sequence will first wear Lens 2 (nelfilcon A), then wear Lens 3 (nesofilcon A) second and then wear Lens 1 (etafilcon A) third .
  Interventions: Device: Lens 1 (etafilcon A); Device: Lens 2 (nelfilcon A); Device: Lens 3 (nesofilcon A)
- Lens 2 / Lens 1/ Lens 3 (Active Comparator): Each subject will be randomly assigned to one of six unique sequences. Subjects randomized to this sequence will first wear Lens 2 (nelfilcon A), then wear Lens 1 (etafilcon A) second and then wear Lens 3 (nesofilcon A) third. Each lens type will be worn for approximately 2 weeks (12 +/- 2 days).
  Interventions: Device: Lens 1 (etafilcon A); Device: Lens 2 (nelfilcon A); Device: Lens 3 (nesofilcon A)
- Lens 3 / Lens 1 / Lens 2 (Active Comparator): Each subject will be randomly assigned to one of six unique sequences. Subjects randomized to this sequence will first wear Lens 3 (nesofilcon A), then wear Lens 1 (etafilcon A) second and then wear Lens 3 (nelfilcon A) third.
  Interventions: Device: Lens 1 (etafilcon A); Device: Lens 2 (nelfilcon A); Device: Lens 3 (nesofilcon A)
- Lens 3 / Lens 2 / Lens 1 (Active Comparator): Each subject will be randomly assigned to one of six unique sequences. Subjects randomized to this sequence will first wear Lens 3 (nesofilcon A), then wear Lens 2 (nelfilcon A) second and then wear Lens 3 (etafilcon A) third.
  Interventions: Device: Lens 1 (etafilcon A); Device: Lens 2 (nelfilcon A); Device: Lens 3 (nesofilcon A)

INTERVENTIONS:
Device: Lens 1 (etafilcon A) — Each lens type will be worn for approximately 2 weeks (12 +/- 2 days).
  Other Names: 1-Day Acuvue® Moist®
Device: Lens 2 (nelfilcon A) — Each lens type will be worn for approximately 2 weeks (12 +/- 2 days).
  Other Names: Dailies® AquaComfort Plus®
Device: Lens 3 (nesofilcon A) — Each lens type will be worn for approximately 2 weeks (12 +/- 2 days).
  Other Names: Biotrue ONEday

SUMMARY:
This is a single-site, 8-visit, double-masked, cross-over study involving three marketed products as study lenses. Participants will be randomly assigned each lens type, which will be worn for approximately two weeks (12 +/- 2 days) each. Participants will undergo a minimum washout period of 3 days before entering the study and undergo a minimum 7 day washout period between dispensing each lens type.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form;
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol;
* The subject must be willing and able to follow instructions and maintain the appointment schedule;
* The subject must be between the age of 18 and 40 years (inclusive);
* The subject's vertex corrected spherical equivalent distance refraction must be in the range of -0.50 Diopters (D) to -6.00 D in each eye (inclusive);
* The subject's refractive cylinder must not exceed -1.25 Diopters of Cylinder (DC) in each eye after vertexing to the corneal plane;
* The subject must have best corrected visual acuity of 0.2 Logarithm of the Minimum Angle of Resolution (logMAR) or better in each eye;
* The subject must be a current wearer of spherical, soft contact lenses (no toric, bifocal or multifocal contact lenses, no extended wear or monovision) for at least 5 days/week and at least 8 hours/day during the month prior to enrollment;
* The subject must own a wearable pair of spectacles and wear them the day of the initial visit;
* The subject must be an existing wearer of spherical, soft contact lenses in both eyes;
* The subject must have normal eyes (i.e., no ocular medications or infections of any type);
* The subject must be willing to wear the study lenses for a minimum eight hours per day.

Exclusion Criteria:

* Any ocular or systemic allergies or diseases that may interfere with contact lens wear (at the investigator's discretion);
* Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear (at the investigator's discretion);
* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued);
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease;
* Any active ocular infection;
* Is using any topical medications (excluding artificial tears (ATS)) up to two weeks prior to the screening visit;
* Any participants whose habitual contact lenses are used as an extended wear regimen;
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry;
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.);
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear; or clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear;
* Any known hypersensitivity or allergic reaction to the study products;
* Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment;
* Employee or family member of the Centre for Contact Lens Research (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2016-01-18 (Actual); Study Completion 2016-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 78 subjects were enrolled in this study. Of the enrolled subjects 74 subjects were dispensed at least 1 study lens and 4 subjects did not meet the eligbility criteria. Of the dispensed subjects 72 completed the study and 2 subjects were discontinued.
Groups:
- Etafilcon A/ Nelfilcon A/ Nesofilcon A: All subjects that were randomized to receive the etafilcon A lens first, the nelfilcon A lens second and the nesofilcon A lens third.
- Etafilcon A/ Nesofilcon A/ Nelfilcon A: All subjects that were randomized to receive the etafilcon A lens first, the nesofilcon A lens second and the nelfilcon A lens third.
- Nelfilcon A/ Nesofilcon A/ Etafilcon A: All subjects that were randomized to receive the nelfilcon A lens first, the nesofilcon A lens second and the etafilcon A lens third.
- Nelfilcon A/ Etafilcon A/ Nesofilcon A: All subjects that were randomzied to receive the nelfilcon A lens first, the etafilcon A lens second and the nesofilcon A lens third.
- Nesolfilcon A/ Etafilcon A/ Nelfilcon A: All subjects that were randomized to receive the nesofilcon A lens first, the etafilcon A lens second and the nelfilcon A lens third.
- Nesofilcon A/ Nelfilcon A/Etafilcon A: All subjects that were randomized to receive the nesofilcon A lens first, the nelfilcon A lens second and the etafilcon A lens third.
Period: Period 1
Arm/Group | Etafilcon A/ Nelfilcon A/ Nesofilcon A | Etafilcon A/ Nesofilcon A/ Nelfilcon A | Nelfilcon A/ Nesofilcon A/ Etafilcon A | Nelfilcon A/ Etafilcon A/ Nesofilcon A | Nesolfilcon A/ Etafilcon A/ Nelfilcon A | Nesofilcon A/ Nelfilcon A/Etafilcon A
Started | 13 | 12 | 13 | 12 | 12 | 12
Completed | 13 | 12 | 13 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Etafilcon A/ Nelfilcon A/ Nesofilcon A | Etafilcon A/ Nesofilcon A/ Nelfilcon A | Nelfilcon A/ Nesofilcon A/ Etafilcon A | Nelfilcon A/ Etafilcon A/ Nesofilcon A | Nesolfilcon A/ Etafilcon A/ Nelfilcon A | Nesofilcon A/ Nelfilcon A/Etafilcon A
Started | 13 | 12 | 13 | 12 | 12 | 12
Completed | 13 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | Etafilcon A/ Nelfilcon A/ Nesofilcon A | Etafilcon A/ Nesofilcon A/ Nelfilcon A | Nelfilcon A/ Nesofilcon A/ Etafilcon A | Nelfilcon A/ Etafilcon A/ Nesofilcon A | Nesolfilcon A/ Etafilcon A/ Nelfilcon A | Nesofilcon A/ Nelfilcon A/Etafilcon A
Started | 13 | 12 | 12 | 12 | 12 | 12
Completed | 13 | 12 | 12 | 12 | 11 | 12
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Unstatisfactory Lens fitting | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least 1 study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least 1 study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.3 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 25
  White | 45
  Other | 3
Region of Enrollment [Number; unit: Participants]
  North America | 74

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Clue comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2- Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Etafilcon A: All subjects that wore the etafilcon A lens during any one of the 3 periods in the study.
- Nelfilcon A: All subjects that wore the nelfilcon A lens in any of the 3 periods of the study.
- Nesofilcon A: All subjects that wore the nesofilcon A lens in any of the 3 periods in the study.
Arm/Group | Etafilcon A | Nelfilcon A | Nesofilcon A
Number analyzed (Participants) | 72 | 72 | 72
Units on a scale | 58.74 (25.350) | 48.14 (25.166) | 57.32 (25.84)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 6 weeks per subject.
Arm/Group | Etafilcon A | Nelfilcon A | Nesofilcon A
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74 | 0/74

LIMITATIONS AND CAVEATS:
Caution of interpretation of results: A significant first-order carryover effect was noted in the study analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days